CLINICAL TRIAL: NCT03584997
Title: Alveolar Ridge Preservation In Mandibular Molars Using Mixture Of Anorganic Bovine Bone(ABB) And Autogenous Particulate VS Mixture Of Injectable Platelets Rich Fibrin, ABB And Autogenous Particulates (Sticky Bone).
Brief Title: Ridge Preservation In Mandibular Molars Using Mixture Of ABB And Autogenous Particulate VS Sticky Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Darwish Elsayed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5050
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Alveolar Bone Loss; Bone Graft Failure; Alveolar Bone Resorption
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF , ABB & Autogenous Particulate (Experimental): Platelets rich fibrin + anorganic bovine bone + autogenous particulate graft
  Interventions: Procedure: PRF, ABB & Autogenous Particulate
- ABB And Autogenous Particulate (Active Comparator): anorganic bovine bone +autogenous particulate graft
  Interventions: Procedure: ABB And Autogenous Particulate

INTERVENTIONS:
Procedure: ABB And Autogenous Particulate — Mixing the autogenous bone graft aquired at the time of surgery with a 50:50 ration of anorganic bovine bone and filling the socket
  Arms: ABB And Autogenous Particulate
Procedure: PRF, ABB & Autogenous Particulate — adding an injectable platelets rich fibrin to a Mixture of autogenous bone graft aquired at the time of surgery with a 50:50 ration of anorganic bovine bone and filling the socket
  Arms: PRF , ABB & Autogenous Particulate

SUMMARY:
Histological Measurement Comparing the density of the new bone formed during socket preservation technique using a Mixture of Anorganic Bovine Bone(ABB) And Autogenous Particulate vs a Mixture of Injectable Platelets Rich Fibers, ABB And Autogenous Particulates (sticky bone). radiographical measurements of the amount of bone dimensions changes in socket preservation technique in 6-month period using a Mixture Of Anorganic Bovine Bone(ABB) And Autogenous Particulate vs a Mixture Of Injectable Platelets Rich Fibers, ABB And Autogenous Particulates (sticky bone)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hopeless mandibular molars indicated for extraction and implant placement in two stages that indicate socket preservation.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual bony Walls after extraction.
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.
* Patients that refuse to be called back for implant placement post extraction.
* Patients that have exceeded bone resorption surrounding the tooth prior to extraction and require guided bone regeneration.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
histomorphometrical bone quality | 6 month
  histological bone quality measured from a core sample taken from the grafted site

SECONDARY OUTCOMES:
marginal bone loss | 6 month
  alveolar margin bone loss measured be CBCT

IPD SHARING:
Plan to Share IPD: Undecided